CLINICAL TRIAL: NCT03055975
Title: Prevalence and Phenotype of Oral Enterococcus Faecalis
Brief Title: Prevalence of Bacteria Following Endodontic Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Federico Foschi, Dr, King's College London
Other Study IDs: 05/Q0705/051
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Root Canal Infection
Keywords: Bacteria; Root canal treatment; Endodontics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary treatments: Patients undergoing primary root canal treatments. Only teeth which have not previously been accessed are included in this cohort.The source population are adults aged 18-65, referred by their general dental practitioner into specialist endodontic clinics of Guy's Hospital
  Interventions: Diagnostic Test: Detection of residual vital bacteria in the root canal space
- Re-treatments: Patients undergoing re-treatments. Only teeth which had a previous root canal treatment which failed are included in this cohort.The source population are adults aged 18-65, referred by their general dental practitioner into specialist endodontic clinics of Guy's Hospital
  Interventions: Diagnostic Test: Detection of residual vital bacteria in the root canal space

INTERVENTIONS:
Diagnostic Test: Detection of residual vital bacteria in the root canal space — Detection of residual vital bacteria in the root canal space. No intervention, as it is an observational study. Vital bacteria are looked for in the samples taken from the root canal space.
  Other Names: Detection of root canal infection

SUMMARY:
Sampling of accessed root canals with endodontic paper points during treatment and immediately pre-obturation of endodontic root canals was carried out.

DETAILED DESCRIPTION:
Following ethical approval (REC ref: 05/Q0705/051), informed consent was obtained from patients undergoing root canal treatment.The teeth included in the study had been referred to a specialist centre for the treatment of endodontic infection. They all responded negatively to vitality tests and presented pre-operative apical radiolucencies. The source population were referred by their general dental practitioner into specialist endodontic clinics of Guy's Hospital, King's College London Dental Institute.Treatments on the teeth were carried out by a total of 19 postgraduate endodontic students.

ELIGIBILITY:
Inclusion Criteria:

* Patients with single or multi-rooted teeth undergoing root canal treatment.

Exclusion Criteria:

* For certain aspects of the study secondary treatments and vital teeth are excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population are adults aged 18-65, referred by their general dental practitioner into specialist endodontic clinics of Guy's Hospital, King's College London Dental Institute. Both single- and multi-rooted non-vital teeth are included in the study
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-01-30 (Actual); Primary Completion 2017-05-30 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
Detection of residual bacteria during and post root canal treatment | June 2016
  Using a vital fluorescent stain bacteria sampled from the root canal space were detected during and post root canal treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Foschi, Dr, Principal Investigator — King's College London
Locations (1):
- King's College London, Dental Institute, Floor 22, Endodontics, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
IPD is not planned to be made available to other researchers as of yet

REFERENCES:
- [Derived] Herzog DB, Hosny NA, Niazi SA, Koller G, Cook RJ, Foschi F, Watson TF, Mannocci F, Festy F. Rapid Bacterial Detection during Endodontic Treatment. J Dent Res. 2017 Jun;96(6):626-632. doi: 10.1177/0022034517691723. Epub 2017 Feb 1. PMID 28530469